CLINICAL TRIAL: NCT02420990
Title: Randomized Comparison of Evidence-Based Protocols for Adolescents With ADHD in Specialty Care: Behavioral Only Versus Integrated Behavioral and Medication Interventions
Brief Title: Integrated Treatment for Adolescents With ADHD
Acronym: CASALEAP IT2A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCORI-1403-13704
Record Dates: First submitted 2015-03-27; First posted 2015-04-20 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: ADHD; Substance Use Disorders
Keywords: ADHD; Adolescents; Substance Use Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Only- Treatment (Active Comparator): All participants will receive behavioral interventions (CASH-AA): family psycho-education in ADHD symptoms, executive functioning, and developmental impacts; family-based motivation and ADHD accommodation interventions; and academic training focused on home environment support and organizational skills.
  Interventions: Behavioral: Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)
- Integrated Treatment (Experimental): Half of the participants will also receive medication decision-making interventions (MIP): ADHD medication psychoeducation, family decision-making interventions, and (for those who elect to start medication) coordinated medication management.
  Interventions: Behavioral: Medication Integration Protocol (MIP); Behavioral: Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)

INTERVENTIONS:
Behavioral: Medication Integration Protocol (MIP)
  Arms: Integrated Treatment
Behavioral: Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) exists in 20-50% of the 3 million adolescents annually enrolled in outpatient mental health and substance use treatment. Adolescents with ADHD present deficits in attention, self-regulation, and social competence that significantly impede achievement of developmental and educational milestones. Currently there are only two evidence-based treatment options for this age group: academic training and stimulant medications. Both options remain vastly underutilized. Academic training is not available in most school settings and rarely implemented in clinical care. Similarly, ADHD medications are rarely utilized with adolescents in primary or specialty care for a host of reasons related to stigma, misinformation about effects and side effects, and adolescent autonomy issues. Moreover, the widespread fragmentation of pharmacological versus behavioral services prevents families from making informed treatment selections.

The primary objective of this randomized parametric trial is to compare the effectiveness of behavioral only versus integrated (behavioral plus medication decision-making) interventions for adolescents with ADHD in outpatient behavioral services. The behavioral intervention, Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA), contains three components: ADHD psychoeducation, family-based motivational interventions, and academic training. The medication decision-making intervention, Medication Integration Protocol (MIP), contain three components: psychoeducation about ADHD medication, family decision-making, and medication management. The study will compare the effects of two legitimate treatment options for adolescents with ADHD on service utilization, behavioral symptoms, and quality of life. It will generate new evidence on patient-centered treatment selection that aligns with family-specific principles and treatment goals.

This parametric comparative trial will randomly assign 140 inner-city adolescents with ADHD to (1) CASH-AA Only or (2) CASH-AA + MIP. Treatment will occur in community behavioral health clinics. All participants will receive behavioral interventions (CASH-AA): family psychoeducation in ADHD symptoms, executive functioning, and developmental impacts; family-based motivation and ADHD accommodation interventions; and academic training focused on home environment support and organizational skills. Half of the participants will also receive medication decision-making interventions (MIP): ADHD medication psychoeducation, family decision-making interventions, and (for those who elect to start medication) coordinated medication management. Half of the sample will have comorbid substance use problems. Treatment will occur in three community clinics; therapists will be randomly assigned to study condition. Caregivers and adolescents will complete assessments at baseline, 3, 6, and 12-month follow-up. Multilevel modeling will compare the effectiveness of each condition on key patient and service use outcomes. Patient-centered analyses will explore differential treatment effects based on (a) Medication decision (yes/no); (b) Substance use comorbidity (yes/no); (c) Race/Ethnicity (Hispanic, African American).

Quantitative outcome analyses will test for service use effects, symptom reduction, and quality of life improvements that are primary reasons for seeking clinical services. Qualitative interviews will document family-specific rationale for decisions about medication, compliance with behavioral and medication interventions, and suggestions for improving services and service integration. Note that families assigned to CASH-AA Only will retain the option of pursuing ADHD medication through treatment-as-usual procedures at their respective clinic. Similarly, families assigned to CASH-AA + MIP will not be required to start ADHD medication. Instead, they will receive informed-choice interventions and can choose when and if to start medication; the study will assess the impact of these decisions on clinical outcomes.

If proven efficacious, the CASH-AA and MIP protocols could be rapidly disseminated individually or as an integrated protocol into routine behavioral healthcare settings. The protocols can also be readily combined with other behavioral treatments to form a multicomponent treatment package for adolescents with co-occurring behavior problems. In addition, the family-based, patient-centered CASH-AA and MIP protocols could be delivered in conjunction with other family-based treatments or with individual approaches that flexibly include caregivers in multiple treatment sessions. This makes CASH-AA and MIP highly efficient clinical resources for addressing ADHD-related problems in any outpatient setting that serves adolescents and their families.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver able to participate in treatment
* Adolescent meets DSM-5 diagnostic criteria for ADHD
* Adolescents who are substance users (50% of sample) meet ASAM criteria for non-intensive outpatient services
* Adolescent not enrolled in any other behavioral treatment
* Caregiver expresses desire, and adolescent expresses willingness, to participate in outpatient treatment
* Family has health benefits that meet the requirements of study treatment sites, all of which accept a broad range of insurance plans including Medicaid.

Exclusion Criteria:

* Intellectual Disability or Autism-Spectrum Disorder
* Medical/psychiatric illness requiring hospitalization
* Current psychotic symptoms; active suicidal ideation
* Severe substance use problems that require immediate relief (detox or residential placement)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Hogue, Ph.D., Principal Investigator — Director of Adolescent and Family Research
Locations (1):
- The National Center on Addiction and Substance Abuse at Columbia University, New York, New York, United States

REFERENCES:
- [Background] Hogue A, Bobek M, Tau GZ, Levin FR. Clinical Strategies for Integrating Medication Interventions Into Behavioral Treatment for Adolescent ADHD: The Medication Integration Protocol. Child Fam Behav Ther. 2014 Oct 1;36(4):280-304. doi: 10.1080/07317107.2014.967631. PMID 25505817
- [Background] Hogue A, Bobek M, Evans SW. Changing Academic Support in the Home for Adolescents with Attention-Deficit/Hyperactivity Disorder: A Family-Based Clinical Protocol for Improving School Performance. Cogn Behav Pract. 2016 Feb;23(1):14-30. doi: 10.1016/j.cbpra.2014.07.002. Epub 2014 Jul 25. PMID 34103882
- [Derived] Hogue A, Horan Fisher J, Dauber S, Bobek M, Porter N, Henderson CE, Evans SW. Randomized Trial of Academic Training and Medication Decision-Making for Adolescents with ADHD in Usual Care. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):874-887. doi: 10.1080/15374416.2020.1716362. Epub 2020 Feb 20. PMID 32078394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 partnering treatment clinics from March 2015 to February 2018.
Groups:
- Behavioral Only- Treatment: All participants will receive behavioral interventions (CASH-AA): family psycho-education in ADHD symptoms, executive functioning, and developmental impacts; family-based motivation and ADHD accommodation interventions; and academic training focused on home environment support and organizational skills.
  Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)
- Integrated Treatment: Half of the participants will also receive medication decision-making interventions (MIP): ADHD medication psychoeducation, family decision-making interventions, and (for those who elect to start medication) coordinated medication management.
  Medication Integration Protocol (MIP)
  Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)
Period: Baseline
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Started | 53 | 92
Completed | 53 | 92
Not Completed | 0 | 0
Period: 3-Month Follow-up
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Started | 53 | 92
Completed | 53 | 92
Not Completed | 0 | 0
Period: 6-Month Follow-up
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Started | 53 | 92
Completed | 53 | 92
Not Completed | 0 | 0
Period: 12-Month Follow-up
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Started | 53 | 92
Completed | 53 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Integrated Treatment: About half of the participants will also receive medication decision-making interventions (MIP): ADHD medication psychoeducation, family decision-making interventions, and (for those who elect to start medication) coordinated medication management.
  Medication Integration Protocol (MIP)
  Changing Academic Support in the Home for Adolescents with ADHD (CASH-AA)
- Total: Total of all reporting groups
Arm/Group | Behavioral Only- Treatment | Integrated Treatment | Total
Number analyzed (Participants) | 53 | 92 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 91 | 144
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.03 (1.84) | 14.68 (1.99) | 14.79 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 32 | 41
  Male | 44 | 60 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 39 | 60
  Not Hispanic or Latino | 32 | 52 | 84
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 15 | 22
  White | 25 | 36 | 61
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 19 | 34 | 53
Region of Enrollment [Number; unit: participants]
  United States | 53 | 92 | 145

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptoms: ADHD Symptoms (Inattention, Hyperactivity/Impulsivity) and Comorbid Problems (Conduct and Mood Problems, Substance Use).
Description: ADHD Symptoms were assessed using the Mini International Neuropsychiatric Interview (Version 5.0). A count of symptoms (range 0-14) was utilized with higher numbers represent more symptoms.
  Delinquency was assessed using the National Youth Survey Self-Report Delinquency Scale (SRD). A count of delinquent acts was utilized (range 0-68) with higher numbers represent more delinquent acts.
  Substance Use was captured with the Comprehensive Addiction Severity Index for Adolescents. Total score was utilized (range 0-60) with higher numbers represent greater substance use.
  Externalizing and Internalizing Symptoms were measured with the Child Behavior Checklist. Higher scores correspond to more symptoms; scores on each item range from 0 to 2, and the study variable was calculated by summing items within each scale (externalizing scale range = 0 - 62 units on a scale; internalizing scale range = 0-64 units on a scale).
Time Frame: Baseline to One Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Number analyzed (Participants) | 53 | 92
units on a scale
  ADHD Symptoms- Inattentive | 6.42 (2.43) | 6.90 (2.43)
  ADHD Symptoms- Hyperactive | 3.23 (2.60) | 4.00 (3.18)
  Delinquent Acts | 13.75 (31.03) | 5.15 (8.99)
  Internalizing Symptoms | 10.20 (8.83) | 9.31 (8.32)
  Externalizing Symptoms | 16.30 (11.45) | 16.76 (12.91)
Statistical Analysis 1: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Latent Growth Curve Modeling; Slope = -.31
Statistical Analysis 2: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Latent Growth Curve Modeling; Slope = -.67
Statistical Analysis 3: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; p = 0.05, Latent Growth Curve Modeling; Slope = .05
Statistical Analysis 4: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; p = 0.05, Latent Growth Curve Modeling; Slope = .56
Statistical Analysis 5: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; p = 0.05, Latent Growth Curve Modeling; Slope = -.72

2. Primary Outcome: Change From Baseline in Quality of Life. Improvements in Executive Functioning and School Functioning.
Description: Executive Functioning was measured with two subscales (self-regulation and self-organization) of the Behavior Rating Inventory of Executive Function. Higher scores correspond to greater difficulty with behavior regulation and organization; scores on each item range from 0 to 2, and the study variable was calculated by summing the scores in each scale (23 items per scale; range 0-46 per scale).
  School Functioning was measured three ways:
  Self-report grades which was coded to reflect 1=Mostly As, 2=As and Bs, 3=Mostly Bs, 4=Bs and Cs, 5=Mostly Cs.
  Academic Self-Efficacy was measured using four dichotomous items from the Motivated Strategies for Learning Questionnaire, 1 = endorsing self-efficacy, 0 = no self-efficacy (range =0-4).
  Homework problems checklist. Higher scores indicate more problems with homework; scores on each item range from 0 to 3; the study variable was calculated by summing the 11 scale items (total score range = 0-33).
Time Frame: Baseline to One Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Number analyzed (Participants) | 53 | 92
units on a scale
  Self-regulation | 48.81 (12.36) | 50.94 (12.98)
  Self-organization | 25.40 (5.81) | 26.04 (5.82)
  Grades | 4.35 (1.50) | 4.50 (1.60)
  Academic Self-Efficacy | .10 (.85) | -.04 (.78)
  Homework Problems | 14.95 (9.57) | 14.84 (9.38)
Statistical Analysis 1: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Linear Growth Curve Modeling; Slope = -1.78
Statistical Analysis 2: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Latent Growth Curve Modeling; Slope = -.64
Statistical Analysis 3: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Linear Growth Curve Modeling; Slope = .07
Statistical Analysis 4: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Latent Growth Curve Modeling; Slope = .00
Statistical Analysis 5: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; Latent Growth Curve Modeling; Slope = -1.44

3. Primary Outcome: Treatment Attendance.
Description: Treatment Attendance [sum of the total number of individual, family, and group sessions attended] and Medication Management Sessions [total number of sessions attended] were collected from agency records. Medication Use, coded as "1 = on" or "0 = off" medication at each follow-up point, was captured with the Services Assessment for Children and Adolescents
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: Sessions
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
Number analyzed (Participants) | 53 | 92
Sessions | 12.8 (11.4) | 19.4 (14.3)
Statistical Analysis 1: Comparison: Behavioral Only- Treatment vs Integrated Treatment; Test type: Superiority; p = .56, Regression, Linear; Mean Difference (Final Values) = 6.6

ADVERSE EVENTS:
Time Frame: Each participant was monitored from baseline interview through 1 year follow-up.
Arm/Group | Behavioral Only- Treatment | Integrated Treatment
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/92
Other Adverse Events (participants affected / at risk) | 0/53 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02420990/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02420990/ICF_001.pdf